CLINICAL TRIAL: NCT01692990
Title: Study on the Effect of Fish Oil and Appetite
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AAstrup (Other)
Responsible Party: Sponsor-Investigator, AAstrup, Associate Professore Lotte Lauritzen, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LL-spec1
Record Dates: First submitted 2012-05-14; First posted 2012-09-26 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-09

CONDITIONS: Obesity; Cachexia
Keywords: Appetite; Fish oil; Long-chain n-3 fatty acids
MeSH Terms: conditions — Obesity; Cachexia | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental): 5 g/d in 10 capsules, providing 3.5 g of long-chain n-3 fatty acids
  Interventions: Dietary Supplement: Fish oil
- Soy bean oil (Placebo Comparator): 5 g/d in 10 capsules
  Interventions: Dietary Supplement: Fish oil

INTERVENTIONS:
Dietary Supplement: Fish oil — For 3 weeks 5 g/d in 10 capsules, providing 3.5 g long-chain n-3 fatty acids in the fish oil period. Cross-over between arms with 1 week of wash out

SUMMARY:
20 normal-weight healthy subjects (10 males, 10 females) were in two periods given 10 of 0.5-mL capsules/day of fish oil and soybean oil for 3 weeks. In the end of each period they were given a standard breakfast and asked to report their appetite on visual analogue scales (VAS) immediately before and after the meal. The results were analyzed in accordance with the paired design under consideration of both supplement sequence and gender.

DETAILED DESCRIPTION:
In a randomized cross-over design, 20 normal-weight healthy subjects (10 males, 10 females) were given 10 of 0.5-mL capsules/day of fish oil and soybean oil for 3 weeks. In the end of each period they were given a standard breakfast and asked to report their appetite on visual analogue scales (VAS) immediately before and after the meal. The results were analyzed in accordance with the paired design under consideration of both supplement sequence and gender.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (18.5<BMI<25 kg/m2).
* Healthy.

Exclusion Criteria:

* Subjects taking medication that could influence appetite.
* Subjects with special nutritional needs e.g. pregnant and lactating, seriously ill or old people.
* Subjects that had had fish oil-supplements for four weeks prior to the intervention period.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Appetite and satiation | October 7th - November 25th 2011
  Appetite and satiation were measured by visual analogue scales (VAS), which assessed satiation, hunger, fullness and desire to eat. Each scale was 100 mm in length with words anchored at each end, expressing the most positive and negative rating of each category.

SECONDARY OUTCOMES:
Weight change | October 7th - November 25th 2011
  Body weight was measured on the same scale without shoes and wearing light clothing in the morning before breakfast.

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Lauritzen, PhD, Principal Investigator — Department of Human Nutrition
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark